CLINICAL TRIAL: NCT01922908
Title: SAfety of Mesenchymal Stromal Cells for Ischemic Stroke
Brief Title: Mesenchymal Stromal Cells for Ischemic Stroke
Acronym: SAMCIS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Plan to change the trial design
Sponsor: Sean Savitz (Other)
Responsible Party: Sponsor-Investigator, Sean Savitz, Professor, Department of Neurology, Director, Stroke Program, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAMCIS
Record Dates: First submitted 2013-08-06; First posted 2013-08-14 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Ischemic Stroke
Keywords: Ischemic; Stroke; Stem Cells; MSC; Allogeneic; Bone Marrow
MeSH Terms: conditions — Ischemic Stroke; Ischemia; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSC infusion (Active Comparator): Allogeneic bone marrow derived mesenchymal stem cells given in one dose 3-10 days after stroke symptom onset
  Interventions: Biological: MSC Infusion
- SHAM infusion (Placebo Comparator): Infusion of normal saline placebo
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: MSC Infusion — Allogeneic bone marrow derived mesenchymal stem cells given in one dose 3-10 days after stroke symptom onset
  Arms: MSC infusion
Biological: Placebo Comparator — Normal saline
  Arms: SHAM infusion

SUMMARY:
The purpose of this study is to determine if mesenchymal stem cells given by IV is feasible and safe in patients with recent ischemic stroke and to decide the maximum tolerated dose when given between 3-10 days after an ischemic stroke.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study. . Approximately 48 subjects will be enrolled in the trial, undergo a real or SHAM MSC IV infusion and will be follow out to 1 year. There will potentially be 4 Cohorts with the dose escalation at a 3:1 randomization schedule

Objectives:

* The primary hypothesis' are that intravenous administration of allogeneic bone marrow derived mesenchymal stem cells is feasible and safe in patients with recent ischemic stroke and to determine the maximum tolerated dose (MTD) of IV MSCs when administered sub-acutely between 3-10 days following ischemic stroke.
* The secondary hypothesis is that allogeneic MSC transplantation will improve functional outcome after recent ischemic stroke.

Safety and clinical efficacy points to be evaluated at Day 7 clinic visit, Day 30, Day 60, Day 90, and Day 180. Primary outcome or Primary endpoint of the study is to define the safety or harm of the MSCs

ELIGIBILITY:
Inclusion Criteria:

1. acute ischemic stroke
2. age 18 to 83 years
3. post stroke mRS > 3
4. NIHSS of 7-25
5. Deficits on the total NIHSS can be lower than 7 provided the patients have moderate aphasia or visual loss (2 on the Best Language or Visual loss NIHSS subcomponent) *Criteria for mRS not used for this category of subjects
6. Last seen normal st within 3-9 days prior to stroke. Time of onset for wake-up stroke will be defined as the time the patient woke up with symptoms.
7. stem cell transplantation procedure must be performed between 3-10 days after stroke symptom onset

Exclusion Criteria:

1. Ischemic stroke, primary hemorrhagic or traumatic lesion of the brain or myocardial infarction within past 30 days prior to current stroke.
2. Mechanical heart valve
3. Uncontrolled seizure disorder, defined as a seizure within the last 6 months
4. Developmental delay
5. Chronic kidney disease
6. Hepatic disease or altered liver function
7. Pulmonary disease
8. Cancer within 5 years prior to study
9. Prior immunosuppression, including chemotherapy within last 3 years
10. Known HIV
11. Uncorrected coagulopathy or severe anemia
12. Pregnancy
13. Unable to undergo MRI or CT scan
14. Imaging shows clinically significant hemorrhage

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of IV MSCs | 24 hours

SECONDARY OUTCOMES:
Improved functional outcome | 1 year
  as assessed by changes in mRS, NIHSS, Fugyl-Meyer and Barthel Index

CONTACTS AND LOCATIONS:
Overall Officials: Sean Savitz, MD, Principal Investigator — The University of Texas Health Science Center, Houston